CLINICAL TRIAL: NCT00992056
Title: Comparative Effects of Nebivolol Versus Metoprolol on Sodium Sensitivity and Renal Sodium Handling in Hypertensive Hispanic Postmenopausal Women
Brief Title: Nebivolol Versus Metoprolol: Sodium Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Richard A. Preston, Chief, Division of Clinical Pharmacology, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20090654
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoprolol/Nebivolol (Experimental): Metoprolol/Nebivolol: Metoprolol 50 mg titrated to 100 mg then nebivolol 5 mg titrated to 10 mg
  Interventions: Drug: nebivolol; Drug: Metoprolol
- Nebivolol/Metoprolol (Experimental): Metoprolol 50 mg titrated to 100 mg then Nebivolol 5 mg titrated to 10 mg
  Interventions: Drug: nebivolol; Drug: Metoprolol

INTERVENTIONS:
Drug: nebivolol — 5 mg titrated to 10 mg daily versus matching placebo
  Other Names: Bystolic
Drug: Metoprolol — Metoprolol 50 mg titrated to 100 mg
  Other Names: Toprol

SUMMARY:
Research objectives

The objective of this randomized, placebo-controlled, 2 period crossover clinical trial is to determine the effects of nebivolol versus metoprolol on ambulatory blood pressure, the blood pressure response to dietary sodium loading, and renal handling of an acute sodium load in postmenopausal women with hypertension.

Hypothesis

Nebivolol will result in a blunted response of blood pressure to oral sodium administration and improved renal handling of an intravenous sodium load in comparison with metoprolol in hypertensive postmenopausal women.

Research plan

Study design

The study consisted of a randomized crossover trial of the effects on sodium sensitivity and renal sodium handling of nebivolol versus metoprolol. All study procedures were carried out under the direct supervision of the Principal Investigator in the outpatient and inpatient research unit of the University of Miami Division of Clinical Pharmacology.

Primary endpoint

Change in 24-hour mean systolic blood pressure determined by 24-hour ambulatory blood pressure monitor (ABPM) from the final day of low sodium to the final day of high sodium in nebivolol versus metoprolol

DETAILED DESCRIPTION:
This investigation consisted of a randomized, open-label, 2-Treatment Period (metoprolol versus nebivolol) crossover clinical trial conducted in postmenopausal women with stage 1 hypertension. Nineteen of 24 participants completed all phases of the protocol and had 4 technically adequate ABPM determinations.

Each randomized 4-week Treatment Period was with either nebivolol 5 mg daily titrated to 10 mg daily versus metoprolol 50 mg daily increased to 100 mg. Participants were randomly assigned in blocks of 2 to either arm of the crossover trial: Metoprolol/Nebivolol or Nebivolol/Metoprolol.

Participants returned at weekly (7 days ± 4 days) intervals during all outpatient study phases. On the day of a scheduled visit, participants were instructed not to take their medication at home, but to bring the medication with them to the visit. Participant visits were scheduled in the morning and all evaluations were performed at drug trough (24 ± 2 hours after the previous day's dose). Medications for that day were administered after all evaluations planned for that visit had been completed. At each visit participants were questioned directly about compliance and any missed or delayed doses. In addition pill counts were conducted at each visit.

Eleven-day Inpatient Confinement Period Both 4-week outpatient Treatment Periods were followed by an 11-day inpatient confinement period in the clinical pharmacology research unit (CPRU). During Days 1-5 participants received a diet designed to contain approximately 30 mmol Na and 50 mmol K. On Day 5 a determination of 24-hour ABPM was performed while continuing to receive this low sodium diet. During Days 6-10 participants received a diet designed to contain approximately 200 mmol Na and 50 mmol K. On Day 10 of this high sodium period ABPM was performed while the subjects continued to receive the 200 mmol Na and 50 mmol K diet. The response to increased dietary sodium was defined as the difference between the ABPM measurements conducted on Day 5 and Day 10. On day 11 a sodium handling study was performed to determine the effects of nebivolol versus metoprolol on sodium excretion (UnaV) following 1 liter 0.9% saline administered over 2 hours. All meals were designed with the supervision of a certified dietitian, provided by the University of Miami Hospital Food Service, and directly supervised by CPRU staff.

Renal sodium handling following a 1 L saline challenge. On Day 11 of the inpatient confinement period, while continuing to receive the 200 mmol Na 50 mmol K diet, an intravenous saline load test was performed. Beginning at approximately 0600, baseline urine for sodium, potassium, and creatinine was collected for two hours. At the midpoint of this 2-hour urine collection, blood was taken for sodium, potassium, and creatinine. At approximately 0800 1 L 0.9% normal saline was infused over 2 hours. Urine collections were performed hourly for six one-hour periods for sodium, potassium, and creatinine. Hour 1 and 2 collections were during the saline infusion. Hour 3-6 collections were post saline infusion. Blood pressure and heart rate were determined at baseline and at each hour during the collection period.

At hour 1 midpoint (30 minutes after the infusion was started), and the midpoint of each hourly urine collection for a total of 6 collection periods, blood was taken for creatinine, sodium, and potassium. Immediately following the 6 one-hour collection periods, the subject resumed the standard diet. Meals were identical and served at the same time on Day 11 for both periods. Urine was then collected and volume recorded at intervals of 6-8 hours, 8-12 hours and 12-24 hours. Aliquots were sent for creatinine, sodium, and potassium.

Nebivolol was provided in 5, 10 and 20 mg tablets by Forest Laboratories, New York, New York. Metoprolol ER was purchased as the generic product in 25, 50 and 100 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Women > 45 years of age.
2. Self-identified as Hispanic ethnicity.
3. Have hypertension defined as:

   * Systolic blood pressure 140-159 mm Hg off antihypertensive medications
   * Diastolic 90-99 mm Hg off antihypertensive medications
4. Blood pressure will be calculated as the mean of 3 consecutive office cuff measurements at rest (sitting). In order to be eligible for treatment, subjects must meet the above definition of hypertension at screening visits off antihypertensive medications
5. Natural menopause at least 1 year (no menstruation for 1 year) prior to screening or had a bilateral oophorectomy at least 3 months prior to study participation.
6. No clinically significant or unstable coexisting medical condition in the estimation of the study PI
7. No clinically significant abnormalities of physical exam or laboratory data in the estimation of the PI
8. Concomitant medications will be evaluated on a case by case basis by the study PI
9. Renal function as assessed by a Cockcroft-Gault estimated glomerular filtration rate (GFR) of >70 ml/min
10. Signed informed consent and the ability to understand the study and its procedures

Exclusion Criteria:

1. Inability to understand the study or provide informed consent
2. History of adverse effects or intolerance to nebivolol or beta-blockers
3. Previous treatment with nebivolol within the preceding six months.
4. Significant or unstable cardiovascular, pulmonary, renal, gastrointestinal, hepatic, endocrine, or central nervous system as determined by the principal investigator.
5. Clinically significant abnormalities of physical examination or laboratory data as determined by the principal investigator.
6. The subject has donated or lost more than 450 mL of blood or has received transfusion of any blood or blood products within 30 days prior to screening.
7. Receiving treatment with diuretics, non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, steroids, or other agents known to influence blood pressure, renal function, or sodium sensitivity. Any concomitant medications will be reviewed by the study PI on a case-by-case basis. In general, no concomitant medication is preferred. Any medication may be tapered/discontinued with consent of patient and at the discretion of the study PI.
8. Grapefruit and Seville oranges are not allowed at any time during the study.
9. Any disease or condition that, in the opinion of the investigator, could compromise the absorption, accumulation, metabolism, or excretion of the study medication.
10. Current alcohol or drug abuse.
11. Smoking of more than 10 cigarettes per day.

Min Age: 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Preston, MD MSPH MBA, Principal Investigator — University of Miami
Locations (1):
- Division of Clinical Pharmacology Clinical Pharmacology Research Unit (CPRU) 1500 NW 12th Ave 15-West., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nebivolol/Metoprolol: Nebivolol 5 mg titrated to 10 mg then Metoprolol 50mg titrated to 100 mg.
- Metoprolol/Nebivolol: Metoprolol 50 mg titrated to 100 mg then nebivolol 5 mg titrated to 10 mg
Period: Treatment Period 1 (6 Weeks)
Arm/Group | Nebivolol/Metoprolol | Metoprolol/Nebivolol
Started | 12 | 12
Completed | 11 (February 2012) | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Washout Period (2 Weeks)
Arm/Group | Nebivolol/Metoprolol | Metoprolol/Nebivolol
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Treatment Period 2 (6 Weeks)
Arm/Group | Nebivolol/Metoprolol | Metoprolol/Nebivolol
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nebivolol/Metoprolol: Nebivolol 5 mg titrated to 10 mg then Metoprolol 50 mg titrated to 100 mg
- Total: Total of all reporting groups
Arm/Group | Metoprolol/Nebivolol | Nebivolol/Metoprolol | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Mean Systolic Blood Pressure by ABPM From Day 5 of Low Sodium to Day 10 of High Sodium
Time Frame: Day 5, Day 10
Population: 24 subjects were randomized. Three withdrew informed consent during the study. One was withdrawn during the washout period. One completed all phases of the study but had a faulty ABPM reading on the last determination
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Metoprolol: Participants who received Metoprolol 50 mg daily increased to 100 mg daily. If goal blood pressure (<140/<90 mmHg) was not achieved at week 3, the metoprolol was titrated to 200 mg.
- Nebivolol: Participants who received Nebivolol 5 mg daily increased to 10 mg daily. If goal blood pressure (<140/<90 mmHg) was not achieved at week 3, the metoprolol was titrated to 20 mg.
Arm/Group | Metoprolol | Nebivolol
Number analyzed (Participants) | 19 | 19
mmHg | 7.7 [3.1 to 12.3] | 9.3 [4.6 to 13.9]

ADVERSE EVENTS:
Arm/Group | Metoprolol | Nebivolol
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol (N=24) | Nebivolol (N=24)
Redness in eyes (Eye disorders) | 2 (2) | 0 (0) — Symptoms occurred in both subjects during metoprolol
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Symtoms occurred during metoprolol
Common cold symptoms (Infections and infestations) | 0 (0) | 1 (1) — Symptoms occurred during nebivolol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No